CLINICAL TRIAL: NCT04353011
Title: Psychological Impact of Quarantine in Chronic Pain Patient During COVID-19 Outbreak
Acronym: DolPsyCOVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_45; 2020-A00912-37 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-05

CONDITIONS: Sars-CoV2; Chronic Pain
Keywords: Psychological impact; COVID-19
MeSH Terms: conditions — Chronic Pain; COVID-19

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with chronic painful
  Interventions: Other: questionnaire assesment

INTERVENTIONS:
Other: questionnaire assesment — questionnaire assesment

SUMMARY:
In the context of quarantine with COVID-19, we will study the experience and psychological impact of pain in adult patients living with chronic pain. We will evaluate the link between the question of physical and psychological confinement in the experience of pain in this particular situation

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic pain
* Patient in confinement
* Patient with sufficient understanding of the French language

Exclusion Criteria:

* Non adult patient
* patient without quarantine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patient will be interviewed par internet questionnaire (patient association / AFVD)
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale questionnaire | 1 week from baseline on

SECONDARY OUTCOMES:
Quality of life (SF36) | 1 week from baseline on
self-reported questionnaire for painful | 1 week from baseline on
qualitive questionnaire | 1 week from baseline on

CONTACTS AND LOCATIONS:
Overall Officials: Anne BERA, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France